CLINICAL TRIAL: NCT01541475
Title: Neuroimaging Study of Bupropion Treatment in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, In Kyoon Lyoo, Professor, Ewha Womans University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 112063; GSK IIT
Record Dates: First submitted 2012-02-17; First posted 2012-03-01 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Bupropion; Escitalopram

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escitalopram + Bupropion (Experimental)
  Interventions: Drug: Bupropion, Escitalopram
- Escitalopram (Active Comparator)
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Bupropion, Escitalopram — Week 0-1: Escitalopram 10mg, Bupropion 150mg Week 2-3: Escitalopram 10mg, Bupropion 300mg Week 4-8: Escitalopram 20mg, Bupropion 300mg
  Arms: Escitalopram + Bupropion
Drug: Escitalopram — Week 0-3: Escitalopram 10mg Week 4-8: Escitalopram 20mg
  Arms: Escitalopram

SUMMARY:
The current study is being conducted in patients with major depression. The study aims to 1) investigate the combined effects of selective serotonin reuptake inhibitor (SSRI) and bupropion compared to SSRI alone on the improvements of depressive symptoms, fatigue, hypersomnia, and neurocognitive functions, 2) observe structural/functional/chemical changes using magnetic resonance imaging (MRI), 3) and examine a relationship between the improvements of depressive symptoms, fatigue, and hypersomnia and the neural changes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 65
* Diagnosis of major depressive disorder (MDD) as assessed by the Structured Clinical Interview for DSM-IV (SCID-IV)
* Individuals who provided written consent for participation.

Exclusion Criteria:

* Presence of any major physical or neurological illness (e.g., head trauma, epilepsy, seizure, stroke, cerebral tumor, multiple sclerosis, cerebrovascular disease, narrow-angle glaucoma, drug hypersensitivity, etc.)
* Diagnosis of any Axis I disorder other than MDD or presence of symptoms requiring hospitalization
* Intelligence quotient (IQ) below 80
* Contraindications to magnetic resonance imaging (e.g., pacemaker implantation, claustrophobia, etc.)
* Unstable medical illness or other abnormalities observed at the screening or laboratory tests
* Women who are pregnant, breastfeeding, or planning pregnancy
* Allergy or tolerance to the clinical trial medication
* Presence of any physical illness that contraindicates the clinical trial medication (e.g., epilepsy, history of uncontrollable narrow-angle glaucoma)
* Use of psychoactive medications that may affect brain imaging findings

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Depressive Symptom Scores at 8 Weeks | Baseline and at 8 Weeks
Change from Baseline in Depressive Symptom Scores at 4 Weeks | Baseline and at 4 Weeks
Change from Baseline in Depressive Symptom Scores at 1 Week | Baseline and at 1 Week

SECONDARY OUTCOMES:
Number of Participants with Adverse Events | 1 Week
Change from Baseline in Neurocognitive Function as Expressed as Z Scores Transformed Using the Control Group Mean and Distribution Values at 8 Weeks | Baseline and 8 Weeks
Changes from Baseline in Brain Structure and Function, Analyzed Using the Computational Approach | Baseline and 8 Weeks
Number of Participants with Adverse Events | 4 Weeks
Number of Participants with Adverse Events | 8 Weeks
Changes in Fatigue Severity Scale scores | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: In Kyoon Lyoo, MD, PhD, MMS, Principal Investigator — Ehwa W. univ hospital
Locations (1):
- Seoul National University Hospital, Biomedical Research Institute, Seoul, Seoul, South Korea